CLINICAL TRIAL: NCT07230964
Title: Early Feasibility Study of the Correlation Between an Impedance Cardiography Test for Decompensation and the Development of Left Ventricular Replacement Fibrosis
Brief Title: Correlation Between an Impedance Cardiography Test for Decompensation and the Development of Left Ventricular Replacement Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dermed Diagnostics, Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: ICG Decompensation LV Fibrosis
Record Dates: First submitted 2025-11-09; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
Keywords: impedance cardiography; decompensation; aortic stenosis; fibrosis; myocardial replacement fibrosis
MeSH Terms: conditions — Aortic Valve Stenosis; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Impedance cardiography test (Experimental): The ICG upright/supine test, using the HYPERGRAPH, will be used to show the difference in the compensatory response between normal LV function and decompensation in HF.
  Interventions: Device: Impedance Cardiography Upright/Supine Test

INTERVENTIONS:
Device: Impedance Cardiography Upright/Supine Test — This ICG upright/supine test is a comparison of [dZ/dt]max in the supine position to [dZ/dt]max in an upright position for assessing decompensation.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of impedance cardiography (ICG), the HYPERGRAPH test, in detecting left ventricular decompensation in patients with aortic stenosis, compared to cardiac magnetic resonance (CMR) imaging findings. The study aims to obtain usable ICG test data on six patients with aortic stenosis who have recently undergone CMR scans with late gadolinium enhancement, and who do not have a history of myocardial infarction or cardiac amyloidosis. The hypothesis to be tested is that the HYPERGRAPH can accurately detect left ventricular decompensation associated with replacement fibrosis obtained from CMR imaging.

DETAILED DESCRIPTION:
BACKGROUND:

The decision to perform transcatheter aortic valve replacement (TAVR) often occurs after there is permanent heart damage. Therefore, there is a need for a novel method of identifying patients with less than severe aortic stenosis who are at imminent risk of heart damage. The concept is that the onset of left ventricular (LV) decompensation is the tipping point that marks the loss of cardiac reserve and the formation of myocardial fibrosis. This is an observational study to gather data pertaining to the possible link between a simple noninvasive test using impedance cardiography (ICG) to detect LV decompensation in patients with moderate aortic stenosis and the development of LV replacement fibrosis. Valvular heart disease (VHD) is a common cause of heart failure (HF). Aortic stenosis, one of the most serious and common forms of VHD, is characterized both by progressive valve narrowing and the LV remodeling response. Moderate aortic stenosis (moderate leaflet calcification) is in Stage B of the American College of Cardiologists (ACC)/American Heart Association (AHA) guidelines for the management of VHD, which specify maximum aortic velocity less than 4.0 m/s or mean aortic pressure gradient less than 40 mmHg, and no symptoms. In fact, some aortic stenosis patients with those valve hemodynamics have symptoms. Also, patients with the same valve characteristics can have very different LV functions ranging from normal myocardium to LV decompensation with significant replacement fibrosis. This suggests that only considering the characteristics of the valve, without looking for LV dysfunction, may be insufficient for determining an appropriate time for TAVR. Currently, commercially available valves are indicated for severe calcific aortic stenosis in patients with symptomatic VHD. This is Stage D in the ACC/AHA VHD guidelines which specify valve hemodynamics of maximum aortic velocity ≥ 4.0 m/s or mean aortic gradient ≥ 40 mmHg. However, clinical studies show that often the decision for TAVR is after there is significant heart damage. This suggests that early intervention, when appropriate, could reduce all-cause mortality and improve outcomes compared with conservative management. In other words, an appropriate time for TAVR could be prior to Stage D. The dilemma is that, even with symptoms, the heart team lacks a clear indication to proceed with TAVR when the maximum aortic velocity is less than 4.0 m/s and the mean aortic gradient is less than 40 mmHg. The shortcoming of watchful waiting is the increased risk of mortality. The common symptoms for aortic stenosis are angina, syncope, and dyspnea. The most serious symptom is dyspnea, which is associated with congestive HF. From the onset of overt dyspnea, 50% of the patients are dead within 2 years. Even patients with the least serious symptom of angina have a mortality rate of 50% within 5 years of the onset of the angina. Myocardial Fibrosis: Myocardial fibrosis is the key pathological feature associated with LV remodeling during the transition from hypertrophy to HF. Myocardial fibrosis can be divided into diffuse fibrosis, which occurs earlier and is reversible, and replacement fibrosis, which occurs later and is irreversible. In theory, an appropriate time for TAVR would be prior to formation of replacement fibrosis. Diffuse and replacement fibrosis in the myocardium are increased with aortic stenosis but are only weakly associated with the severity of valve narrowing. In fact, patients with moderate aortic stenosis can have normal myocardium, diffuse fibrosis, or replacement fibrosis. Gap in Current Knowledge: LV remodeling due to aortic stenosis cannot be accurately predicted from the degree of valve narrowing alone and should be assessed independently. Detection of subclinical LV decompensation potentially could be helpful in assessing the progression of fibrosis associated with the transition from hypertrophy to HF. The ICG test described in this study is a potential candidate for the needed simple and inexpensive method of detecting LV decompensation.

Impedance Cardiography:

The ICG technology has been available for over 50 years. ICG was initially commercialized to noninvasively monitor cardiac output. The capability of the technology expanded to include assessment of the hemodynamic function of the cardiovascular system in HF. ICG has been used to detect decompensation in patients with heart failure, but ICG has not been used specifically to detect decompensation in patients with moderate aortic stenosis. This is a new clinical application where the onset of decompensation could be important. Gathering data on ICG readings in the upright and supine positions for detecting decompensation in patients with aortic stenosis is the purpose of this project. The scientific basis of the technology is the following. The resistance to flow of an alternating electrical current is known as impedance, and the tissue resistance to an applied current is termed electrical bioimpedance (Z). An electric field within the thorax is created by applying alternating, high frequency, low-amplitude current from a constant-current source via a set of electrocardiograph-type electrodes on the neck and abdomen. The real-time impedance signal resembles the aortic pressure wave. To facilitate intuitive interpretation, the signal is inverted so that a decrease in impedance appears as a rise in the displayed waveform. It is known that the rate of pressure rise in the ascending aorta, dP/dt (which is the slope of the upstroke of the pressure wave during the ejection phase), is an indication of contractility. During systole, the aortic pressure change (which is the cause) directly correlates with the impedance change (which is the result). The differentiated impedance signal, dZ/dt, correlates directly with dP/dt. On the dZ/dt waveform, the ejection wave is defined as the portion of the dZ/dt waveform during ventricular ejection. The highest point on the ejection wave is [dZ/dt]max, measured in ohms per second. In systole, the major source of the impedance change is blood movement in the aorta. The height of the ejection wave, [dZ/dt]max, correlates with left ventricular contractility.

Novel Method of Assessing Decompensation: The ground truth behind the ICG upright/supine test is Starling's law of the heart. For ventricular function, the Frank-Starling relation states that the force of ventricular contraction is affected by the end-diastolic length of the fibers comprising the myocardial wall, which is closely related to the end-diastolic volume. Body position affects the distribution of blood volume. End-diastolic volume is influenced by the distribution of blood volume between the intrathoracic and extrathoracic compartments. When a person is upright, the gravitational force causes blood to pool in lower portions of the body which increases extrathoracic blood volume at the expense of intrathoracic blood volume. For a person at rest, the maneuver of changing posture from upright to supine causes a decrease in extrathoracic blood volume and an increase in intrathoracic blood volume. This increases venous return to the heart (preload) and end-diastolic volume. In a heart which remains compensated, the contractile force increases as muscle length increases. An increase in LV end-diastolic volume causes the muscle to stretch within its elastic limit and results in a greater contractile force. In other words, in compensation, supine [dZ/dt]max is greater than upright [dZ/dt]max. [29] The Frank-Starling curve represents the stress/strain relationship of ventricular performance (LV stress) to LV end-diastolic volume (LV strain). In a normal heart, the curve is ascending, indicating that an increase in end-diastolic volume results in an increase in contractile force. In HF, the left ventricle becomes decompensated. The onset of decompensation, represented by the plateau of the heart failure curve, occurs when the left ventricle has no more cardiac reserve. This is the tipping point when the LV myocardium is stretched to its elastic limit. The onset of decompensation is indicated by the upright [dZ/dt]max being the same as the supine [dZ/dt]max. In theory, the onset of decompensation marks the beginning of the replacement of viable myocardial tissue with fibrotic non-contractile tissue. The descending part of the HF curve represents worsening decompensation, when the LV myocardium is stretched beyond its elastic limit resulting in a weaker contraction. The weaker the contraction, the slower the blood is ejected from the left ventricle into the aorta. This causes a slower rise (lower slope) of the upstroke of the aortic pressure wave. This is indicated by a smaller value of [dZ/dt]max. As decompensation worsens, the supine dZ/dt]max continues to decrease below the upright [dZ/dt]max. In decompensation, a pathophysiologic alteration is the inability of the heart to move all the blood that is returned from the circulatory system, when a patient is not upright, leading to a buildup of blood to the heart (congestion). The onset of decompensation could be considered the "canary in the coal mine", because it serves as an early warning that the transition from hypertrophy to HF is imminent. Potentially, the onset of LV decompensation could indicate the start of the timing window for considering TAVR for patients with aortic stenosis. Relevant Preliminary Data: For comparisons of LV systolic function across patients, the measure of [dZ/dt]max is normalized by dividing the [dZ/dt]max value by the base impedance (the average electrical bioimpedance) of the thorax (Zo). This is similar to the way that stroke volume is normalized by dividing the stroke volume value by body surface area to produce stroke index. This normalized ICG indicator of LV contractile force is called systolic amplitude (SA). The formula for SA is [dZ/dt]max (in Ω per second) divided by Zo (in Ω). [33] For assessing the compensatory response to postural change, the criterion for a normal compensatory response is upright SA less than supine SA. Decompensation is defined as upright SA ≥ supine SA, indicating that the left ventricle has lost contractile reserve and is performing contrary to normal function according to Starling's law of the heart. The onset of decompensation occurs when upright SA equals supine SA.

Expected Outcome:

The shift from compensation to decompensation could be an important milestone in LV remodeling. In theory, the ICG detected onset of decompensation is a harbinger of the development of LV replacement fibrosis. The expected outcome of this study is a negative ICG test for decompensation in a moderate aortic stenosis patient with a CMR scan.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female at least 18 years of age.

  * No prior history of myocardial infarction or cardiac amyloidosis.
  * Recent CMR scan with late gadolinium enhancement or scheduled for CMR scan with late gadolinium enhancement.
  * A history of:
  * Moderate aortic stenosis and no replacement fibrosis OR Moderate aortic stenosis and symptoms who has replacement fibrosis OR Severe aortic stenosis with replacement fibrosis prior to aortic valve replacement.
  * Able to comprehend and provide informed consent in English.
  * Participants must have intact, healthy skin at the electrode application sites.

Exclusion Criteria:

* • Under 18 years of age

  * Pregnant or breastfeeding women
  * Unable to consent
  * Prisoners
  * History of myocardial infarction
  * History of cardiac amyloidosis
  * Patients with any metal or implant such as IUD, braces, metal fragments implants in the eye, pacemakers (especially Minute Ventilation pacemakers with the MV function activated) defibrillators, or any other electronic cardiac implant.
  * Claustrophobic or afraid or small places.
  * Severe obesity (BMI > 40) that impairs accurate ICG measurement due to difficulties in electrode placement or excessive impedance.
  * Active skin conditions, such as rashes, open wound or significant skin sensitivity at the electrode placement sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between ICG decompensation detection and replacement fibrosis measured by CMR scan | The assessment for each participant will be performed immediately following the one-time ICG test and CMR scan.
  Look for a negative ICG test for decompensation correlating with a CMR scan indicating a very low extracellular volume and a positive ICG test for decompensation correlating with a CMR scan indicating a very high extracellular volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeMarzo AP. Using impedance cardiography with postural change to stratify patients with hypertension. Ther Adv Cardiovasc Dis. 2011 Jun;5(3):139-48. doi: 10.1177/1753944711406770. Epub 2011 Apr 28. PMID 21527444